CLINICAL TRIAL: NCT05874076
Title: The Effects of Mutation on Short Term Physiotherapy Success in Hospitalized COVID-19 Patients: a Prospective Study
Brief Title: Physiotherapy in Mutated COVID-19 Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Giresun University (Other)
Responsible Party: Principal Investigator, Ulkukezbansahin, Head of therapy and rehabilitation department, Giresun University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023
Record Dates: First submitted 2023-05-22; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: COVID-19 Pandemic
MeSH Terms: conditions — COVID-19 | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Covid-19 group (Active Comparator): This group underwent physiotherapy consisting of mobilization, normal range of motion, and a respiratory exercise program.
  Interventions: Behavioral: Physiotherapy
- Mutation group (Experimental): This group underwent physiotherapy consisting of mobilization, normal range of motion, and a respiratory exercise program.
  Interventions: Behavioral: Physiotherapy

INTERVENTIONS:
Behavioral: Physiotherapy — Physiotherapy

SUMMARY:
The prospective study was conducted at a single location within the COVID-19 department of a city hospital. The study included COVID-19 patients who were hospitalized in the COVID-19 service and consulted for physiotherapy, were between the ages of 18 and 65, and had the capacity and inclination to participate in one daily physiotherapy session five days per week.

DETAILED DESCRIPTION:
A hospital's COVID-19 service recruited 32 participants for the study. Patients were divided into two groups: COVID-19 (n=16; age = 53.81 9.48) and mutation (n=16; age = 55.25 10.12). Both groups underwent physiotherapy consisting of mobilization, normal range of motion, and a respiratory exercise program (COVID-19 group: 9.945.85 days; mutation group: 7.632.83 days). Every patient participated in a once-daily physiotherapy program. The patients' muscle strength, mobility, daily activities, exercise capacity, and perception of fatigue were assessed. To compare groups, the mixed repeated measures ANOVA model was used.

ELIGIBILITY:
Inclusion Criteria:

Patients with COVID-19 who were hospitalized in the COVID-19 service Patients were consulted for physiotherapy Patients with the capacity and willingness to participate in one daily physiotherapy session five days a week

Exclusion Criteria:

* Patients who had an exercise contraindication, were uncooperative, had multi-organ failure, had an acute infection, or were PEG-fed were excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
muscle strength | an average of 9 days
  Using a scale developed by the Medical Research Council (MRC), muscle strength was measured. Using this instrument, the muscles of the lower and upper extremities are evaluated bilaterally. Each of the six main muscle groups evaluated receives a score between 0 (no contraction) and 5 (normal contraction).

SECONDARY OUTCOMES:
mobility assessment | an average of 9 days
  For the purpose of measuring mobility, the Rivermead Mobility Index (RMI) was applied.
Exercise capacity | an average of 9 days
  Exercise capacity was evaluated with the 5-repetition sit to stand test (5STS).

CONTACTS AND LOCATIONS:
Overall Officials: ULKU K SAHIN, PhD, Principal Investigator — Giresun University
Locations (2):
- Turkey (Türkiye) (2):
  - Giresun University, Giresun, Gi̇resun
  - Giresun University, Giresun

IPD SHARING:
Plan to Share IPD: No
The datasets generated during and analyzed during the current study are available from the corresponding author on reasonable request.

REFERENCES:
- [Result] Lemhofer C, Gutenbrunner C, Schiller J, Loudovici-Krug D, Best N, Bokel A, Sturm C. Assessment of rehabilitation needs in patients after COVID-19: Development of the COVID-19-rehabilitation needs survey. J Rehabil Med. 2021 Apr 27;53(4):jrm00183. doi: 10.2340/16501977-2818. PMID 33764478
- [Result] Brower RG. Consequences of bed rest. Crit Care Med. 2009 Oct;37(10 Suppl):S422-8. doi: 10.1097/CCM.0b013e3181b6e30a. PMID 20046130
- [Result] Piquet V, Luczak C, Seiler F, Monaury J, Martini A, Ward AB, Gracies JM, Motavasseli D; Covid Rehabilitation Study Group. Do Patients With COVID-19 Benefit from Rehabilitation? Functional Outcomes of the First 100 Patients in a COVID-19 Rehabilitation Unit. Arch Phys Med Rehabil. 2021 Jun;102(6):1067-1074. doi: 10.1016/j.apmr.2021.01.069. Epub 2021 Feb 4. PMID 33548208